CLINICAL TRIAL: NCT04415918
Title: Is Bezlotoxumab Effective, Tolerable and Cost Saving in Preventing Recurrent Clostridium Difficile Infections in Patients With Malignancies? An Exploratory Study
Brief Title: Bezlotoxumab Efficacy and Tolerability in Cancer Patient
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-432
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Clostridium Difficile Infection Recurrence
MeSH Terms: interventions — bezlotoxumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Recruited patient according inclusion/exclusion criteria
  Interventions: Drug: Bezlotoxumab Injection
- Historical control (No Intervention): Cohort of historical patients matched to study population to serve as control

INTERVENTIONS:
Drug: Bezlotoxumab Injection — A single dose of Bezlotoxumab (Zinplava) 10mg/kg (actual body weight) 60-minute intravenous infusion during active CDI treatments.
  Other Names: No intervention
  Arms: Intervention group

SUMMARY:
Investigation of efficacy and tolerability of bezlotoxumab in patients with cancer diagnosis in terms of preventing CDI recurrence.

DETAILED DESCRIPTION:
The study will be prospective, open-label, single center with historical control. All procedures will be conducted according to Good Clinical Practice guidelines and the provisions of the Declaration of Helsinki. Approval of Institutional Review Board at Cooper Health Care will be obtained prior to commencing the study and actively enrolled patients will sign an informed consent form. Data will be collected on a case report form and confidentiality will be protected according to laws and regulations. Study population will include adult cancer patients diagnosed with CDI being treated at MD Anderson cancer center affiliated with Cooper University Hospital, Camden, NJ, USA. The comparison arm will be a historical group of patients treated at the same center with same inclusion/exclusion criteria within the previous 3 years of start date.

Recruited patients will receive a single dose of Bezlotoxumab (Zinplava) 10mg/kg (actual body weight) 60-minute intravenous infusion during active CDI treatments.

For pharmacoeconomic analysis, data collected from the financial department will include total hospitalization costs, drug costs, length of stay, total amount charged and total amount reimbursedpertaining to CDI diagnosis code/ICD-10 for recurrent CDI. The analysis will encompass the perspectives of the hospital and the third party payer. Adjustment of retrospective cost data will be performed using Medical Consumer Price index (MCPI) inflation rates established by Bureau of Labor Statistics. Cost-avoidance analysis will be performed to determine the cost of preventing recurrence. Incremental cost-effectiveness ratio (ICER) defined as the difference in cost divided by difference in outcomes will be reported. The outcome being examined, the percent of recurrences avoided, will be used in the denominator. Graphically, a cost-effectiveness plane will be used to depict the comparison. Secondary analyses will examine specific differences between groups, including total drug costs, length of stay (LOS) and per diem hospitalization costs. Univariate sensitivity analyses will be conducted to determine robustness of the analysis.

Matching of intervention group with control will be based on inclusion/exclusion criteria, sex, and GEIH-CDI propensity score as shown in the table below. Matching will be in the ratio of 1:2. Selected historical control based on inclusion/exclusion criteria will matched to same sex.

Patients treated at MD Anderson cancer center affiliated with Cooper University Hospital Camden, NJ, USA with diagnosis of CDI will be screened using inclusion/exclusion criteria. Eligible patients will be approached for consent. Recruited patients will receive the study intervention either as in-patients or at the out-patient infusion unit according to their current status. The study patients will be followed for 12 weeks (day1 is the day of study intervention) on week1, week2, week 4, week 8 and week 12 (- or + 5 days) until study exit day. Study required clinical data will be collected from medical records on case report form. Financial data will be acquired from accounting department records. Recruited patients will be interviewed on the phone or in person.

Study intervention drug will be stored at the Pharmacy Department, Cooper University Hospital. Shortly before the time of administration, infusion will be prepared as per manufacturer instructions (250 mL infused over 1 hours through 0.22-micron sterile filter controlled by volumetric pump) and transported for administration per the hospital protocol. Patients receiving bezolotoxumab infusion will be under observation and follow up as per study protocol.

To assess recurrence, clinical cure is achieved in patients receiving standard of care treatment and have no diarrhea (< 3 bowel movements per day) for 2 consecutive days following completion of therapy. Patients will be followed by reviewing medical records, in person and by phone.

Tolerability of bezolotoxumab will be assessed by collecting clinical and laboratory data about adverse events as detailed below under adverse experience reporting.

A 10-mL blood sample will be collected from patients in heparinized tubes (processed and/or stored as required by the lab) for genetic DNA profiling. An an assessment of bezlotoxumab efficacy and the correlation with the SNP will be performed.

Withdrawal from the study will be voluntary or at the discretion of investigators/sponsor in case of tolerability concerns, protocol violation or any other reason.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age
2. Diagnosed with any type of malignancy and receiving active treatment (chemotherapy, radiotherapy or biological therapy)
3. Confirmed clinical (patients with unexplained and new-onset >3 unformed stools in 24 hours) and laboratory (a stool toxin test as part of a multistep algorithm) diagnosis of primary or recurrent CDI and receiving standard of care treatment
4. Patient or legally authorized person signs informed consent form -

Exclusion Criteria:

1- Patients with short life expectancy including terminal cancer, multi-organ dysfunction or on compassionate care (as per treating physician) 2- Pregnant or breastfeeding female patients or likely to be pregnant without negative laboratory confirmation 3- Patients with active chronic diarrheal disease 4- Patients with other acute, unstable and life-threatening conditions (acute renal or hepatic failure, sepsis or other severe infections, active bleeding, stroke or myocardial infarction) 5- Patient receiving or planning to receive other CDI interventions like FMT within 3 months of bezlotuxumab therapy 6- Patients who previously received bezlotoxumab within the past 3 months 7- Patients completed active of CDI treatment 8- Patients with any conditions that at discretion of the investigators will compromise patient rights, ability to participate or complete the study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with recurrent CDIs within 12 weeks of initial cure compared with historical group of patients selected with same inclusion/exclusion criteria (same center within 3 years of the start date of the study). | 12 weeks
  Documentation of recurrent CDI infection

SECONDARY OUTCOMES:
Determine if bezlotoxumab infusion add-on treatment is cost saving in patients with malignancies in terms of preventing CDI recurrence. | 12 weeks
  Pharmacoeconomic analysis

OTHER OUTCOMES:
Explore if genetic variants (SNP rs2516513 on xMHC, SNP genotype on IL-8 gene promotor, SNP rs2243250 IL-4 gene,….) are associated with increased recurrence of CDI in this patient population. | 12 weeks
  Genetic analysis is performed to describe gene type

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared